CLINICAL TRIAL: NCT05119075
Title: Unravelling the Impact of Levodopa on Dysfunctional Brain Networks in Parkinson's Disease With Neuropsychiatric Fluctuations
Brief Title: Psychological Effects of Levodopa in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Geneva (Other); Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-01608
Record Dates: First submitted 2021-09-28; First posted 2021-11-12 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Neuropsychiatric fluctuations; Creativity; Shame; Embarrassment; Non-motor symptoms; Hallucinations; Bradyphrenia
MeSH Terms: conditions — Parkinson Disease; Hallucinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dopaminergic ON-drug state first, dopaminergic OFF-drug state second (Experimental): The following examinations and assessments will be performed at visit 3 on regular treatment in dopaminergic ON-drug state and at visit 4 in dopaminergic OFF-drug state (overnight withdrawal of all antiparkinsonian drugs):
  * MRI assessment,
  * Cognitive, neuropsychiatric and neurological assessment,
  * Robot-induced hallucinations through sensorimotor stimulation.
  Interventions: Other: Dopaminergic OFF-drug state; Other: Dopaminergic ON-drug state
- Dopaminergic OFF-drug state first, dopaminergic ON-drug state second (Experimental): The following examinations and assessments will be performed at visit 3 in dopaminergic OFF-drug state (overnight withdrawal of all antiparkinsonian drugs) and at visit 4 on regular treatment in dopaminergic ON-drug state:
  * MRI assessment,
  * Cognitive, neuropsychiatric and neurological assessment,
  * Robot-induced hallucinations through sensorimotor stimulation.
  Interventions: Other: Dopaminergic OFF-drug state; Other: Dopaminergic ON-drug state

INTERVENTIONS:
Other: Dopaminergic OFF-drug state — Dopaminergic OFF-drug state: Overnight withdrawal of dopaminergic antiparkinsonian drugs during visit 3 or 4. The sequence of drug conditions (dopaminergic OFF-drug/ON-drug state or ON-drug/OFF-drug state) will be randomized.
Other: Dopaminergic ON-drug state — Dopaminergic ON-drug state: Patient will be evaluated in his/her regular treatment in dopaminergic ON-drug state at visit 3 or 4. The sequence of drug conditions (dopaminergic OFF-drug/ON-drug state or ON-drug/OFF-drug state) will be randomized.

SUMMARY:
The investigators aim is to study neuropsychiatric symptoms and underlying abnormalities in resting-state fMRI in patients with Parkinson's disease (PD) suffering from neuropsychiatric fluctuations, to enhance the understanding of the pathophysiological mechanisms underlying neuropsychiatric symptoms.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is primarily classified and known as a movement disorder characterized by tremor, bradykinesia and rigidity. However, clinical examination and research have shown that PD extensively affects other systems as well, giving rise to non-motor symptoms (NMS) such as anxiety, sleep disorders, apathy, depression, cognitive impairment, and hallucinations. These non-motor fluctuations (NMF) represent a main source of disability in PD and among those, neuropsychiatric fluctuations are the most frequent. During the dopaminergic OFF-drug state anxiety, apathy, and depression are common, whereas during the dopaminergic ON-drug state euphoria, well-being, impulse control disorders (ICD) and other behavioral addictions, mania, and psychosis might occur.

Despite the severe consequences associated with dopaminergic modulation, the understanding of the pathophysiological mechanisms of neuropsychiatric symptoms is still limited and better detection and more effective treatments are needed. Fluctuating PD is a very powerful model allowing to study opposite psychiatric states intra-individually in both levodopa dopaminergic ON- and OFF-drug state, allowing to abstract many interpersonal variables.

Neurotechnology and advanced neuroimaging techniques can improve the understanding of the neural basis and brain mechanisms of specific neuropsychiatric symptoms in PD. In particular, dynamic functional connectivity (FC) analysis characterizes functional abnormalities from resting state (rs)-fMRI not only in terms of brain activations, but also of whole-brain functional networks and the transitions between maps of activations. The temporal evolution of these networks, assessed with dynamic FC approaches, has recently shown to be relevant in several clinical contexts.

Therefore, the investigators long-term goal is to identify specific resting-state signatures/biomarkers for the individual neuropsychiatric PD symptoms related to disease in dopaminergic OFF-drug state (depression, anxiety, apathy, fatigue, shame, bradyphrenia) and to dopaminergic treatment in dopaminergic ON-drug state (mania, impulse control disorders, hallucinations, psychosis, creative thinking), which might be used in the future as a proxy for the measurement of neuropsychiatric symptoms/fluctuations and thus to assess the effectiveness of specific therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adults above 18 years old
* Male or female
* Diagnosed with Parkinson's disease
* Able to understand instructions, neuropsychological tests and provide written informed consent
* Able to understand the locally used language of the experimental site and speak fluently
* Presence of neuropsychiatric fluctuations, defined as the sum ≥ 3 of items included in the Ardouin Scale of Behaviour in Parkinson's Disease (ASBPD) part 2

Exclusion Criteria:

* Structural brain disease other than Parkinson's disease
* Substance abuse and/or dependence (other than DRT)
* Ongoing depression with suicidal ideation
* Severe tremors/dyskinesia/ interfering with MRI performance
* Participating in a pharmacological study
* Inability to provide informed consent (legal guardianship)
* MRI contraindications
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Correlation of functional connectivity abnormalities with neuropsychiatric fluctuations | ≤ 6 weeks
  Score on the Neuropsychiatric Fluctuations Scale (NFS)
Correlation of functional connectivity abnormalities with shame | ≤ 6 weeks
  Score on the Shame Visual Analogic Scale
Correlation of functional connectivity abnormalities with hallucinations | ≤ 6 weeks
  Score on robot-induced presence hallucination (PH) ratings
Correlation of functional connectivity abnormalities with bradyphrenia | ≤ 6 weeks
  Score on the Bradyphrenia Scale
Correlation of functional connectivity abnormalities with creativity | ≤ 6 weeks
  Score on the Creative Thinking Scale

SECONDARY OUTCOMES:
The role of dopamine on hallucinations | ≤ 6 weeks
  Measurement of the influence of dopamine on hallucinations using the robot-induced presence hallucination (PH) ratings. Assessments will be performed under the two conditions (dopaminergic ON and OFF drug state) and compared. The higher the score, the more hallucinations are experienced by patients.
The role of dopamine on creativity | ≤ 6 weeks
  Measurement of the influence of dopamine on the Creative Thinking Scale. Assessments will be performed under the two conditions (dopaminergic ON and OFF drug state) and compared. The higher the score, the more creative the patients are.
The role of dopamine on shame | ≤ 6 weeks
  Measurement of the influence of dopamine on the Shame Visual Analogic Scale. Assessments will be performed under the two conditions (dopaminergic ON and OFF drug state) and compared. The higher the score, the more shame patients feel.
The role of dopamine on bradyphrenia | ≤ 6 weeks
  Measurement of the influence of dopamine on the bradyphrenia scale. Assessments will be performed under the two conditions (dopaminergic ON and OFF drug state) and compared. The higher the score, the more bradyphrenic the patients are.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Krack, Prof., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (4):
- Switzerland (4):
  - University Hospital Inselspital, Berne, Bern
  - EPFL Campus Biotech, Geneva
  - EPFL Institute of Bioengineering, Geneva
  - University Hospital Geneva (HUG), Geneva

IPD SHARING:
Plan to Share IPD: No